CLINICAL TRIAL: NCT02836782
Title: Dynamics of Viral Reservoir in HIV-positive Patients With or Without HCV Coinfection in the Era of Direct-acting Antiviral and Antiretroviral Drugs
Brief Title: HIV-DNA Dynamics in HIV Monoinfected or HIV/HCV Coinfected Patients
Acronym: ViDyMoCo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Simona Di Giambenedetto, Researcher, Catholic University of the Sacred Heart
Other Study IDs: Prot.7768/16 ID 1086
Record Dates: First submitted 2016-05-05; First posted 2016-07-19 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: HIV
Keywords: HIV/HCV; Antiretroviral therapy; HIV-DNA; Direct acting antiviral

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Naive patients: Patients who begin their first antiretroviral regimen. Blood sample withdrawal
  Interventions: Procedure: Blood sample withdrawal
- Experienced patients: Patients with a history of antiretroviral treatment, switching to a new regimen.
  Blood sample withdrawal
  Interventions: Procedure: Blood sample withdrawal

INTERVENTIONS:
Procedure: Blood sample withdrawal — Blood withdrawal for HIV-DNA or HCV resistance test

SUMMARY:
New markers of viral activity are now under investigation. Aim of the study is to investigate the efficacy of new antiretroviral drugs by monitoring HIV-DNA dynamics in HIV-positive population. In HIV/HCV coinfected population, the study of HIV reservoir dynamics and the analysis of the prevalence of HCV resistance-associated mutations will help clinicians to improve the management of coinfected patients.

DETAILED DESCRIPTION:
New markers of viral activity are now under investigation. Besides HIV-RNA and CD4 cells count, HIV-DNA is an emerging marker of viral reservoir, that seems to be associated with the risk of HIV-related diseases, especially in HCV coinfected patients. New antiretroviral drugs, particularly integrase inhibitors, are expected to decrease residual viremia and, consequently, viral reservoir. Monitoring of HIV-DNA dynamics during antiretroviral treatment could lead to a better management of HIV infected population.

Also, the role of HCV in influencing HIV natural history requires careful monitoring. In particular, with a broader use of direct acting antiretroviral, the analysis of prevalence of HCV resistance associated mutation will be more and more important to manage patients with treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Persons ≥ 18 years-old;
* Signing an informed consent to study participation and data treatment;
* HIV-positive patients, beginning a new antiretroviral treatment patients or with clinically relevant events;
* HCV-positive patients beginning an antiviral treatment with DAA.

Exclusion Criteria:

* Patient's deny
* Clinical contraindications to blood sample withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of HIV-positive patients with a significant HIV-DNA decay after 3 years from a new antiretroviral regimen start | up to 144 weeks

SECONDARY OUTCOMES:
Percentage of HIV/HCV coinfected patients with a significant HIV-DNA decay after 3 years from the enrollment | up to 144 weeks
Measurement of HIV-DNA level during HCV antiviral therapy with DAA in HIV/HCV coinfected patients | up to 24 weeks
Prevalence of HCV resistance-associated variants and their relation with HIV-DNA levels in HIV/HCV coinfected patients, treated or not treated for HCV. | up to 144 weeks
Comparison of the prevalence of HCV resistance-associated variants in HIV/HCV coinfected population versus HCV monoinfected population | up to 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simona Di Giambenedetto, Researcher, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kostrikis LG, Touloumi G, Karanicolas R, Pantazis N, Anastassopoulou C, Karafoulidou A, Goedert JJ, Hatzakis A; Multicenter Hemophilia Cohort Study Group. Quantitation of human immunodeficiency virus type 1 DNA forms with the second template switch in peripheral blood cells predicts disease progression independently of plasma RNA load. J Virol. 2002 Oct;76(20):10099-108. doi: 10.1128/jvi.76.20.10099-10108.2002. PMID 12239284
- [Background] Shiramizu B, Paul R, Williams A, Shikuma C, Watters M, Grove J, Valcour V. HIV proviral DNA associated with decreased neuropsychological function. J Neuropsychiatry Clin Neurosci. 2007 Spring;19(2):157-63. doi: 10.1176/jnp.2007.19.2.157. PMID 17431062
- [Background] Asselah T, Boyer N, Saadoun D, Martinot-Peignoux M, Marcellin P. Direct-acting antivirals for the treatment of hepatitis C virus infection: optimizing current IFN-free treatment and future perspectives. Liver Int. 2016 Jan;36 Suppl 1:47-57. doi: 10.1111/liv.13027. PMID 26725897
- [Background] Bagaglio S, Uberti-Foppa C, Messina E, Merli M, Hasson H, Andolina A, Galli A, Lazzarin A, Morsica G. Distribution of natural resistance to NS3 protease inhibitors in hepatitis C genotype 1a separated into clades 1 and 2 and in genotype 1b of HIV-infected patients. Clin Microbiol Infect. 2016 Apr;22(4):386.e1-386.e3. doi: 10.1016/j.cmi.2015.12.007. Epub 2015 Dec 17. PMID 26706617
- [Background] Di Maio VC, Cento V, Di Paolo D, Aragri M, De Leonardis F, Tontodonati M, Micheli V, Bellocchi MC, Antonucci FP, Bertoli A, Lenci I, Milana M, Gianserra L, Melis M, Di Biagio A, Sarrecchia C, Sarmati L, Landonio S, Francioso S, Lambiase L, Nicolini LA, Marenco S, Nosotti L, Giannelli V, Siciliano M, Romagnoli D, Pellicelli A, Vecchiet J, Magni CF, Babudieri S, Mura MS, Taliani G, Mastroianni C, Vespasiani-Gentilucci U, Romano M, Morisco F, Gasbarrini A, Vullo V, Bruno S, Baiguera C, Pasquazzi C, Tisone G, Picciotto A, Andreoni M, Parruti G, Rizzardini G, Angelico M, Perno CF, Ceccherini-Silberstein F; HCV Italian Resistance Network Study Group. HCV NS3 sequencing as a reliable and clinically useful tool for the assessment of genotype and resistance mutations for clinical samples with different HCV-RNA levels. J Antimicrob Chemother. 2016 Mar;71(3):739-50. doi: 10.1093/jac/dkv403. Epub 2015 Dec 17. PMID 26679249
- [Background] AASLD/IDSA/IAS-USA RETREATMENT OF PERSONS IN WHOM PRIOR THERAPY HAS FAILED. Recommendations for testing, managing, and treating hepatitis C. date accessed 5.01. 2015.
- [Background] Fourati S, Pawlotsky JM. Virologic Tools for HCV Drug Resistance Testing. Viruses. 2015 Dec 4;7(12):6346-59. doi: 10.3390/v7122941. PMID 26690198
- [Background] Perales C, Quer J, Gregori J, Esteban JI, Domingo E. Resistance of Hepatitis C Virus to Inhibitors: Complexity and Clinical Implications. Viruses. 2015 Nov 6;7(11):5746-66. doi: 10.3390/v7112902. PMID 26561827
- [Derived] Lombardi F, Belmonti S, Borghetti A, Fabbiani M, Marchetti S, Tamburrini E, Cauda R, di Giambenedetto S. Evolution of cellular HIV DNA levels in virologically suppressed patients switching to dolutegravir/lamivudine versus maintaining a triple regimen: a prospective, longitudinal, matched, controlled study. J Antimicrob Chemother. 2020 Jun 1;75(6):1599-1603. doi: 10.1093/jac/dkaa058. PMID 32101614